CLINICAL TRIAL: NCT00519168
Title: Sleep, Circadian, Hormonal Dysregulation, and Breast Cancer Survival
Brief Title: Sleep, Circadian Hormonal Dysregulation, and Breast Cancer Survival
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David Spiegel, Jack, Samuel and Lulu Willson Professor in Medicine, Stanford University
Other Study IDs: BRSADJ0013; 97312 (Other: Stanford University Alternate IRB Approval Number); BRSADJ0013 (Other: Stanford University)
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Urinalysis; Phlebotomy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva and blood
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Urine sample — Standard of care
  Other Names: urine test
Device: Electrode sleep recorder — Standard of care
  Other Names: Digital sleep recorder
Procedure: phlebotomy — Standard of care
  Other Names: blood draw

SUMMARY:
Recent research provides evidence that disrupted circadian rhythms, including hormonal patterns and sleep, are associated with increased risk of breast cancer incidence and faster progression to mortality. We have observed that a loss of normal diurnal cortisol rhythm associated with more awakenings during the night predicts early mortality with metastatic breast cancer. Other recent studies have shown that nighttime shift work is associated with higher breast cancer incidence, and in a murine model disrupting circadian cortisol cycles produced a doubling of implanted tumor growth. There is also recent evidence that abnormal clock genes are associated with cancer. However, it is not clear whether sleep disruption per se affects breast cancer progression, or whether such an effect is mediated by hormonal and immune dysregulation of this prevalent and hormone-mediated cancer. We propose to study sleep disruption as a prognostic factor in the progression of metastatic breast cancer. We will also examine sleep patterns in association with disrupted circadian rhythms of cortisol, ACTH, and melatonin as well as measures of immune function known to be salient to breast cancer progression. These are natural killer cell cytoxicity and specific cytokine, IL-6. We plan to recruit 105 women 45 years through 75 years with metastatic or recurrent breast cancer and 20 age and SES-matched controls for a two-week at home sleep study with Actiwatch and two nights of in-home EEG monitoring, followed by 28 hours of continuous blood sampling and one night of EEG sleep monitoring in our lab at Stanford. This will provide a full examination of circadian hormones associated with sleep patterns. We will relate these assessments to the subsequent course of breast cancer progression. Results of this study will provide specific evidence regarding how improved sleep management may affect the course of breast cancer. Aim 1: To study 24-hr diurnal rhythms of HPA axis hormones and melatonin in women with metastatic or recurrent breast cancer. Hypothesis 1: Women with metastatic or recurrent breast cancer will have reduced amplitude and disrupted phase of 24-hr diurnal rhythms of cortisol, ACTH, and melatonin. Aim 2: To describe sleep disruption in women with metastatic breast cancer and examine psychosocial, endocrine, and immune factors that may be associated with sleep disruption. Hypothesis 2: Women with metastatic or recurrent breast cancer will have a higher incidence of both at home and laboratory-examined sleep disruption than control women without breast cancer. Hypothesis 3: Poorer sleep quality will be associated with more pain, more emotional suppression in response to stressors, less emotional support, greater depression and anxiety, and greater perceived and traumatic stress. Hypothesis 4: Poorer sleep quality and quantity of sleep and daytime sleepiness and fatigue will be associated with abnormal circadian neuroendocrine (i.e., cortisol, ACTH, and melatonin) and immune patterns (i.e., suppressed day and night time NK activity and loss of NK rhythms; increased day time IL-6 levels and /or loss of IL-6 rhythm). Aim 3: To study the relationship between sleep disruption and survival time among metastatic and recurrent breast cancer patients. Hypothesis 5: Poorer sleep quality and quantity of sleep will predict shorter survival. Hypothesis 6: Reduced diurnal amplitude and an abnormal phase of cortisol will predict shorter survival. Explanatory Aim 4: To investigate whether sleep disruption mediates the relation of psychosocial factors to health outcomes.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for women with breast cancer:

1. Female
2. Between 45 and 75 years old (45<=>75)
3. Documented metastatic or recurrent breast cancer
4. Karnofsky rating of at least 70% (measure of physical ability used to assess medically ill patients)
5. Residence within the Greater San Francisco Bay Area
6. Proficiency in English sufficient to complete questionnaires
7. Postmenopausal
8. Non smoker (occasional smoking will be ok, they need to agree to stop smoking during study participation. If smoking cessation will cause withdrawal, they can not participate)
9. Willing to go through a 30 day washout period if they are currently on Decadron or any other corticosteroids (depending on the dose, may be able to reduce 30 days to 2 weeks)
10. If taking Benzodiazepines, willing to stop 3 days before the collection of physiological measures, such as the 2 week at home sleep recordings and then the 3 days before and during the GCRC (if not possible, washout period may be reduced to 3 days before and during the CTRU/GCRC stay)
11. Willingness to discontinue taking melatonin one week before the CTRU/GCRC stay
12. Willingness to discontinue any current sleeping medications 3 days before 2 week at home sleep data collection through the end of study participation (if not possible, washout period may be reduced to 3 days before and during the CTRU/GCRC stay)
13. Willingness to abstain from traveling 2 or more time zones away from California (Pacific time), two weeks before and during participation in the study
14. Willing/able to refrain from doing shift-work in a non-traditional schedule (such as 4pm to midnight or 10pm to 6am) starting two weeks before at home sleep collection through the end of study participation.
15. Agree to catheterization for blood sample collection
16. Agrees with the use of heparin during the blood draws (used to keep IV line from clotting)
17. Has graduated high school or obtained GED
18. US Citizen or resident viable for payment, legally

Inclusion criteria for healthy controls:

1. Female
2. Between 45 and 75 years old (45<=>75)
3. No history of any type of cancer
4. Residence within the Greater San Francisco Bay Area
5. Proficiency in English to complete questionnaires
6. Post Menopausal
7. Non-smoker (occasional smoking will be ok, they need to agree to stop smoking during study participation. If smoking cessation will cause withdrawal, they can not participate)
8. If taking benzodiazepines, willing to stop 3 days before the collection of physiological measures, such as the 2 week at home sleep recordings and then the 3 days before and during the GCRC (if not possible, washout period may be reduced to 3 days before and during the CTRU/GCRC stay)
9. Willingness to discontinue taking melatonin one week before the CTRU/GCRC stay
10. Willingness to discontinue any current sleeping medications 3 days before 2 week at home sleep data collection through the end of study participation (if not possible, washout period may be reduced to 3 days before and during the CTRU/GCRC stay)
11. Willingness to abstain from traveling 2 or more time zones away from California (Pacific time), two weeks before and during participation in the study
12. Willing/able to refrain from doing shift-work in a non-traditional schedule (such as 4pm to midnight or 10pm to 6am) starting two weeks before at home sleep collection through the end of study participation
13. Agree to catheterization for blood sample collection
14. Agrees with the use of heparin during the blood draws (used to keep IV line from clotting)
15. Has graduated high school or obtained GED
16. US Citizen or resident viable for payment, legally
17. Pittsburgh Sleep Quality Index (PSQI) score >6

Exclusion Criteria:Exclusion criteria for women with breast cancer:

1. Other active cancers within the past 10 years other than breast cancer, basal cell or squamous cell carcinomas of the skin, or in situ cancer of the cervix
2. Concurrent medical condition likely to influence short term survival (such as liver disease, asthma etc, depending on severity)
3. History of major psychiatric illness that required hospitalization or medication
4. Substance Dependence or abuse
5. Low hematocrit (up to the digression of the PI, may be able to participate in parts of the protocol)
6. Bilateral lymph nodes removed
7. Diagnosis of diabetes (need to check with PI, some mild cases of diabetes may be ok)
8. Positive supraclavicular lymph nodes as the only metastatic lesion at the time of initial diagnosis
9. PICC line too close to the few available veins, viable for catheterization (too high of a risk for infection/complication), and is on the only arm which did not have lymph node surgery

Exclusion criteria for healthy controls:

1. Concurrent medical condition likely to influence short term survival (such as liver disease, asthma etc, depending on severity)
2. History of major psychiatric illness that required hospitalization or medication
3. Substance dependence or abuse
4. Low hematocrit (up to the digression of the PI, may be able to participate in parts of the protocol)
5. Diagnosis of diabetes (need to check with PI, some mild cases of diabetes may be ok)

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2006-09; Primary Completion 2011-08-31 (Actual); Study Completion 2011-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States